CLINICAL TRIAL: NCT01657474
Title: A Prospective, Randomized, Comparative Study of Amniotic Membrane Wound Graft With Weekly Versus BiWeekly Application In the Management of Diabetic Foot Ulcers
Brief Title: Comparative Study of Two Application Regimens of Amniotic Membrane Wound Graft In the Management of Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFDFU002
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

ARMS (2):
- Weekly Application of EpiFix (Experimental): Weekly application of EpiFix plus standard of care
  Interventions: Other: Weekly application of EpiFix plus standard of care
- Biweekly application of EpiFix (Experimental): Biweekly application of EpiFix plus standard of care
  Interventions: Other: Biweekly application of EpiFix plus standard of care

INTERVENTIONS:
Other: Weekly application of EpiFix plus standard of care
  Arms: Weekly Application of EpiFix
Other: Biweekly application of EpiFix plus standard of care
  Arms: Biweekly application of EpiFix

SUMMARY:
The purpose of this study is to determine whether a weekly application of EpiFix human amniotic membrane is more effective than a biweekly application (every two weeks) in the treatment of diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 18 or older
2. Informed consent must be obtained
3. Patient's ulcer must be diabetic in origin and larger than 1cm2. Debridement will be done prior to randomization. Subject's informed consent for participating in this study, must be obtained prior to proceeding with sharp debridement.
4. Patients with Type 1 or Type 2 diabetes (criteria for the diagnosis of diabetes mellitus per ADA).
5. Ulcer must be present for a minimum of four weeks before enrollment/randomization, with documented failure of prior treatment to heal the wound. A two week run in period will precede enrollment/randomization in the trial to document the indolent nature of the wounds selected
6. Additional wounds may be present but not within 3cm of the study wound
7. Wound must be present anatomically on the plantar surface of the foot
8. Patient's ulcer must exhibit no clinical signs of infection.
9. Patient is of legal consenting age.
10. Patient is willing to provide informed consent and is willing to participate in all procedures and follow up evaluations necessary to complete the study.
11. Serum Creatine less then 3.0mg/dl
12. HbA1c less than 12%
13. Patient has adequate circulation to the affected extremity, as demonstrated by one of the following within the past 60 days:

    * Dorsum transcutaneous oxygen test (TcPO2) with results ≥30mmHg, OR
    * ABIs with results of ≥0.7 and ≤1.2, OR
    * Doppler arterial waveforms, which are triphasic or biphasic at the ankle of affected leg

Exclusion Criteria:

1. Patients presenting with an ulcer probing to bone (UT Grade IIIA-D). A positive probe-to-bone will be confirmed when bone or joint can be felt with a sterile, ophthalmological probe.
2. Patients whose index diabetic foot ulcers are greater than 25cm2.
3. Patients considered not in reasonable metabolic control, confirmed by an HbA1c greater than 12% within previous 90 days,
4. Patients whose serum creatinine levels are 3.0mg/dl or greater.
5. Patients with a known history of poor compliance with medical treatments.
6. Patients who have been previously randomized into this study, or are presently participating in another clinical trial
7. Patients who are currently receiving radiation therapy or chemotherapy.
8. Patients with known or suspected local skin malignancy to the index diabetic ulcer.
9. Patients diagnosed with autoimmune connective tissues diseases.
10. Non-revascularizable surgical sites
11. Active infection at site
12. Any pathology that would limit the blood supply and compromise healing;
13. Patients that have received a biomedical or topical growth factor for their wound within the previous 30 days
14. Patient who are pregnant or breast feeding
15. Patient who are taking medications that are considered immune system modulator which could affect graft incorporation.
16. Allergy to Gentamycin or Streptomycin
17. Wounds greater than one year in duration without intermittent healing
18. Wound improving greater than 20% over the first two weeks of the trial using standard of care dressing and Cam Boot

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Mean time to healing | up to 12 Week

SECONDARY OUTCOMES:
Proportion of completely healed ulcers | Week 4 and Week 12
Percent change in wound area | Week 4 and Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Charles M. Zelen, DPM, Principal Investigator — Professional Education and Research Institute
Locations (2):
- United States (2):
  - Professional Education and Research Institute, Roanoke, Virginia
  - Professional Education and Research Institute, Salem, Virginia